CLINICAL TRIAL: NCT00400894
Title: Annexin A3 (ANXA3) as Protein-Based Marker for Non-Invasive Molecular Diagnostics of Prostate Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: ProteoSys AG (Industry)
Collaborators: Charite University, Berlin, Germany (Other); University Hospital Tuebingen (Other); Medical Centre, Ludwigshafen, Germany (Unknown); Medical University Innsbruck (Other)
Other Study IDs: EA 4/033/06
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Last update posted 2007-02-05 (Estimated); Status verified 2007-02

CONDITIONS: Prostate Cancer; Benign Prostatic Hyperplasia; Prostatic Intraepithelial Neoplasia
Keywords: prostate cancer; annexin A3; early detection; exprimate urine
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia; Prostatic Intraepithelial Neoplasia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Emerging from a differential proteomic study of sample pairs of prostate cancer and benign tissue, annexin A3 (ANXA3) was chosen as a potential novel biomarker for the early and non-invasive diagnosis of prostate cancer. We wanted to show or investigate, that:

* ANXA3 can be detected in urine after standard digital rectal examination.
* ANXA3 has better specificities than tPSA, in particular in the grey zone of PSA
* ANXA3 can help avoid unnecessary biopsies
* ANXA3 can in the long run replace PSA as a marker

DETAILED DESCRIPTION:
The aim of this multi centre and double-blinded study was to investigate specificities and sensitivities of early detection of prostate cancer with a new protein biomarker, annexin A3, using urine after digital rectal examination/massage (exprimate urine) in direct comparison to the corresponding measurements of the gold standard, total PSA. The material obtained by this non-invasive procedure was moreover used to determine appropriate cut-off values and optimal fractions (e.g. after centrifugation) and calibrations for quantitative measurements of this novel marker.

Patients (500-750) were (and are) continuously recruited from four clinical centres in Germany (Berlin, Tübingen, Ludwigshafen) and Austria (Innsbruck). The major aspect was:

• Can annexin A3 provide a better specificity than tPSA, in particular in the grey zone of PSA (2-10 ng/ml) and can annexin A3 thus contribute to a significant reduction of invasive transrectal biopsies?

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histological confirmation of adenocarcinoma of the prostate
* Patients with benign prostatic hyperplasia (confirmed by histology of lance biopsies or TUR-P)

Exclusion Criteria:

* Patients with rectal extirpation
* Patients with renal or bladder tumors

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 750
Dates: Start 2005-09; Study Completion 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schostak, PD Dr., Principal Investigator — University Medical Centre Charité, Berlin, Germany; André Schrattenholz, Prof. Dr., Study Director — ProteoSys AG, Mainz, Germany

REFERENCES:
- [Background] Wozny W, Schroer K, Schwall GP, Poznanovic S, Stegmann W, Dietz K, Rogatsch H, Schaefer G, Huebl H, Klocker H, Schrattenholz A, Cahill MA. Differential radioactive quantification of protein abundance ratios between benign and malignant prostate tissues: cancer association of annexin A3. Proteomics. 2007 Jan;7(2):313-22. doi: 10.1002/pmic.200600646. PMID 17205602
- [Derived] Schostak M, Schwall GP, Poznanovic S, Groebe K, Muller M, Messinger D, Miller K, Krause H, Pelzer A, Horninger W, Klocker H, Hennenlotter J, Feyerabend S, Stenzl A, Schrattenholz A. Annexin A3 in urine: a highly specific noninvasive marker for prostate cancer early detection. J Urol. 2009 Jan;181(1):343-53. doi: 10.1016/j.juro.2008.08.119. Epub 2008 Nov 13. PMID 19012935